CLINICAL TRIAL: NCT00173966
Title: A Case Control Study to Investigate the Possible Association Between Atrial Fibrillation and Endothelium Dysfunction by Using Flow-Mediated Vasodilation Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701155
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-12

CONDITIONS: Atrial Fibrillation; Endothelial Function
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Endothelial function is closely related to the hemostasis , vascular tone, and organ perfusion in cardiovascular system, and its dysfunction would cause overactivation of the coagulative system to induce thrombus formation. So we study the relationship between the endothelial function and atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Lone AF patients and normal controls

Exclusion Criteria:

* DM, hypertension, hyperlipidemia, smoking, pregnancy,

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Juey Jen Hwang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan